CLINICAL TRIAL: NCT06129565
Title: The Use of Q-Collar to Increase CSF Drainage in Low-pressure Hydrocephalus Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Participants not enrolled due to interest in the project
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UKansasQcollarLPH
Record Dates: First submitted 2023-10-03; First posted 2023-11-13 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Low Pressure Hydrocephalus
MeSH Terms: conditions — Hydrocephalus, Normal Pressure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Q-collar Intervention (Experimental): All patients with low-pressure hydrocephalus that qualify for the study and agree to participate will receive the Q-collar for intervention
  Interventions: Device: Q-collar

INTERVENTIONS:
Device: Q-collar — Q-collar is placed for all patients that are admitted with low-pressure hydrocephalus

SUMMARY:
The investigators hypothesize that the Q-collar compression on bilateral internal jugular veins of patients with low pressure hydrocephalus will decrease venous drainage from the intracranial space, therefore increasing intracranial volume, decreasing brain compliance, and increasing CSF drainage through the shunt. This should improve persistent hydrocephalus symptoms and demonstrate improved ventricular drainage on imaging with decompressed ventricles.

DETAILED DESCRIPTION:
Low-pressure hydrocephalus is an entity that is rare and difficult to manage. At this institution, Dr. Paul Camarata uses a method of "neck-wrapping" in those low-pressure hydrocephalus patients that were admitted for complications with their shunt, hypothesized to decrease venous outflow from the intracranial space, increase venous pressure within the cranium and therefore increase the turgor in the brain tissue allowing for CSF to more easily be pushed out of the ventricular space and through the drain. This would relieve the hydrocephalus symptoms and reduce ventricular size on imaging. The advent of the Q-collar for reducing TBI in contact sports functions in a similar way to the "neck-wrapping" used at this institution, but via the simplified tool of the collar. It functions by compressing the internal jugular veins bilaterally to increase intracranial volume and prevent "brain slosh" that can occur in contact sports that leads to brain injury. The collar in contrast to the neck wrap occupies a smaller surface area, which the investigators hypothesize will reduce the discomfort that is commonly associated with neck wrap. Furthermore, applying this Q-collar to low pressure hydrocephalus patients that struggle with symptom management while inpatient, the investigators hypothesize that CSF drainage will improve with wearing the collar via increased intracranial volume and lower brain compliance, therefore improving persistent hydrocephalus symptoms that are limiting on patient quality of life.

ELIGIBILITY:
Inclusion Criteria:

* adult with low-pressure hydrocephalus, able to cranial imaging, able to provide consent or have surrogate decision maker that is able to provide it for them

Exclusion Criteria:

* pediatric patients, patients that can't consent or don't have a surrogate decision maker, patients that can't get cranial imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Ventricular drainage | within 4-6 weeks
  Amount of ventricular drainage with Q collar treatment
Ventricular size | within 4-6 weeks
  change in ventricular size with Q collar treatment

SECONDARY OUTCOMES:
Change in low-pressure hydrocephalus symptoms | 4-6 weeks
  Patients surveyed daily regarding low-pressure hydrocephalus symptoms including headache, altered mental status, blurry vision, other. Will document if worse, unchanged, or improved.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smith DW, Bailes JE, Fisher JA, Robles J, Turner RC, Mills JD. Internal jugular vein compression mitigates traumatic axonal injury in a rat model by reducing the intracranial slosh effect. Neurosurgery. 2012 Mar;70(3):740-6. doi: 10.1227/NEU.0b013e318235b991. PMID 21904255
- [Background] Turner RC, Naser ZJ, Bailes JE, Smith DW, Fisher JA, Rosen CL. Effect of slosh mitigation on histologic markers of traumatic brain injury: laboratory investigation. J Neurosurg. 2012 Dec;117(6):1110-8. doi: 10.3171/2012.8.JNS12358. Epub 2012 Sep 21. PMID 22998060
- [Background] Sindelar B, Bailes J, Sherman S, Finan J, Stone J, Lee J, Ahmadian S, Zhou Y, Patel V, Smith D. Effect of Internal Jugular Vein Compression on Intracranial Hemorrhage in a Porcine Controlled Cortical Impact Model. J Neurotrauma. 2017 Apr 15;34(8):1703-1709. doi: 10.1089/neu.2016.4648. Epub 2016 Dec 16. PMID 27573472
- [Background] Mannix R, Morriss NJ, Conley GM, Meehan WP 3rd, Nedder A, Qiu J, Float J, DiCesare CA, Myer GD. Internal Jugular Vein Compression Collar Mitigates Histopathological Alterations after Closed Head Rotational Head Impact in Swine: A Pilot Study. Neuroscience. 2020 Jun 15;437:132-144. doi: 10.1016/j.neuroscience.2020.04.009. Epub 2020 Apr 10. PMID 32283181
- [Background] Myer GD, Yuan W, Barber Foss KD, Thomas S, Smith D, Leach J, Kiefer AW, Dicesare C, Adams J, Gubanich PJ, Kitchen K, Schneider DK, Braswell D, Krueger D, Altaye M. Analysis of head impact exposure and brain microstructure response in a season-long application of a jugular vein compression collar: a prospective, neuroimaging investigation in American football. Br J Sports Med. 2016 Oct;50(20):1276-1285. doi: 10.1136/bjsports-2016-096134. Epub 2016 Jun 15. PMID 27307271
- [Background] Myer GD, Yuan W, Barber Foss KD, Smith D, Altaye M, Reches A, Leach J, Kiefer AW, Khoury JC, Weiss M, Thomas S, Dicesare C, Adams J, Gubanich PJ, Geva A, Clark JF, Meehan WP 3rd, Mihalik JP, Krueger D. The Effects of External Jugular Compression Applied during Head Impact Exposure on Longitudinal Changes in Brain Neuroanatomical and Neurophysiological Biomarkers: A Preliminary Investigation. Front Neurol. 2016 Jun 6;7:74. doi: 10.3389/fneur.2016.00074. eCollection 2016. PMID 27375546
- [Background] Dinsmore M, Hajat Z, Brenna CT, Fisher J, Venkatraghavan L. Effect of a neck collar on brain turgor: a potential role in preventing concussions? Br J Sports Med. 2022 Jun;56(11):605-607. doi: 10.1136/bjsports-2021-103961. Epub 2021 Nov 25. PMID 34824061
- [Background] Filippidis AS, Kalani MY, Nakaji P, Rekate HL. Negative-pressure and low-pressure hydrocephalus: the role of cerebrospinal fluid leaks resulting from surgical approaches to the cranial base. J Neurosurg. 2011 Nov;115(5):1031-7. doi: 10.3171/2011.6.JNS101504. Epub 2011 Jul 29. PMID 21800965
- [Background] Strand A, Balise S, Leung LJ, Durham S. Low-Pressure Hydrocephalus: A Case Report and Review of the Literature. World Neurosurg. 2018 Jan;109:e131-e135. doi: 10.1016/j.wneu.2017.09.120. Epub 2017 Sep 28. PMID 28962963